CLINICAL TRIAL: NCT00871364
Title: Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Actavis Group hf 50 mg Venlafaxine Hydrochloride Tablets and Wyeth Pharmaceuticals (Effexor®) 50 mg Venlafaxine Hydrochloride Tablets
Brief Title: A Relative Bioavailability Study of 50 mg Venlafaxine Hydrochloride Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AA32215
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; venlafaxine; Healthy subjects
MeSH Terms: interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): VENLAFAXINE TABLETS 50 mg, single dose
  Interventions: Drug: VENLAFAXINE TABLETS 50 mg , single dose
- B (Active Comparator): Effexor® (venlafaxine HCl) Tablets equivalent to 50 mg venlafaxine, single dose
  Interventions: Drug: Effexor® Tablets equivalent to 50 mg venlafaxine

INTERVENTIONS:
Drug: VENLAFAXINE TABLETS 50 mg , single dose — A: Experimental Subjects received EMCURE PHARMACEUTICALS LTD. formulated products under fed conditions
  Other Names: venlafaxine
  Arms: A
Drug: Effexor® Tablets equivalent to 50 mg venlafaxine — B: Active comparator Subjects received Wyeth Pharmaceuticals Inc. formulated products under fed conditions
  Other Names: venlafaxine
  Arms: B

SUMMARY:
The purpose of this study to assess the single-dose relative bioavailability of Actavis Group hf 50 mg venlafaxine hydrochloride tablets with Wyeth Pharmaceuticals (Effexor®) 50 mg venlafaxine (as venlafaxine hydrochloride) tablets under fed conditions.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, 2-period, 2-sequence, crossover design.

Official Title: Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Actavis Group hf 50 mg Venlafaxine Hydrochloride Tablets and Wyeth Pharmaceuticals (Effexor®) 50 mg Venlafaxine Hydrochloride Tablets in Healthy Adult Volunteers under Fed Conditions.

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female volunteers, 18-55 years of age.
* Weighing at least 60 kg for males and 52 kg for females and within 15% of their ideal weights (Table of "Desirable Weights of Adults", Metropolitan Life Insurance Company, 1983).
* Medically healthy subjects with clinically normal laboratory profiles, vital signs and ECGs.
* Females of childbearing potential were either sexually inactive (abstinent) for 14 days prior to the first dose, throughout the study and for 6 days following the last dose or were using one of the following acceptable birth control methods:

  * surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) 6 months minimum;
  * IUD in place for at least 3 months;
  * barrier methods (condom, diaphragm) with spermicide for at least 14 days prior to the first dose, throughout the study and for 6 days following the last dose;
  * surgical sterilization of the partner (vasectomy for 6 months minimum);
  * hormonal contraceptives for at least 3 months prior to the first dose of the study and up to 6 days following the last dose. Other birth control methods may have been deemed acceptable. Postmenopausal women with amenorrhea for at least 2 years were eligible.
* Gave voluntary written informed consent to participate in the study.

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, haematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* In addition, history or presence of:

  * alcoholism or drug abuse within the past year;
  * hypersensitivity or idiosyncratic reaction to venlafaxine or other selective serotonin and norepinephrine reuptake inhibitors;
  * glaucoma.
* Female subjects who were pregnant or lactating.
* Subjects who tested positive at screening for HIV, HbsAg or HCV.
* Subjects who received monoamine oxidase (MAO) inhibitors within 28 days prior to dosing.
* Subjects who used any drugs or substances known to be strong inhibitors of CYP enzymes (formerly known as P450 enzymes) within 10 days prior to the first dose.
* Subjects who used any drugs or substances known to be strong inducers of CYP enzymes (formerly known as P450 enzymes) within 28 days prior to the first dose.
* Subjects who donated 50 to 499 mL of blood within 30 days and more than 499 mL within 56 days prior to the first dose.
* Subjects who, through completion of the study, would have donated in excess of:

  * 500 mL of blood in 14 days; or
  * 1500 mL of blood in 180 days; or
  * 2500 mL of blood in 1 year.
* Subjects whose PR interval is >200 msec at screening and prior to dosing.
* Subjects whose QTc interval is >450 msec at screening and prior to dosing.
* Subjects who completed another clinical trial within 28 days prior to the first dose.
* Subjects who were on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-04; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morelli,, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Saint-Laurent, Montreal, Quebec, Canada